CLINICAL TRIAL: NCT03239613
Title: Postoperative Hypofractionated Intensity-modulated Radiation Therapy with Concurrent Chemotherapy in Cervical Cancer: a Prospective Exploratory Trial (POHIM_CCRT Trial)
Brief Title: Postoperative Hypofractionated Intensity-modulated Radiation Therapy with Concurrent Chemotherapy in Cervical Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2017-03-091-003
Record Dates: First submitted 2017-08-02; First posted 2017-08-04 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2023-11

CONDITIONS: Cervix Cancer; Radiotherapy, Adjuvant; Radiotherapy, Intensity-Modulated; Hypofractionated Dose; Chemotherapy, Concurrent
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- POHIM-CCRT (Other): postoperative adjuvant concurrent chemotherapy with hypofractionated IMRT (2.5 Gy/fraction, 16 fractions, once a day)
  Interventions: Other: POHIM-CCRT

INTERVENTIONS:
Other: POHIM-CCRT — postoperative adjuvant concurrent chemotherapy with hypofractionated IMRT (2.5 Gy/fraction, 16 fractions, once a day)

SUMMARY:
To investigate the acute toxicities, late toxicities, and treatment results when the early cervical cancer patients are treated by concurrent chemotherapy with hypofractionated intensity-modulated radiotherapy (2.5 Gy X 16 fractions, once a day) after radical hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed cervical cancer
* radical hysterectomy and pelvic lymph node dissection was done
* histologically indicated adjuvant chemoradiotherapy (more than one as below)

  * positive pelvic lymph node metastasis
  * positive parametrial invasion
  * positive tumor involvement on surgical margin
* ECOG performance status 0 or 1
* Bone marrow function: granulocyte ≥1.0 x 1000/µl, platelet ≥30 x 1000/µl, hemoglobin ≥10 g/dl
* Kidney function: Creatinine <2.0 mg/dL, Bilirubin 1.5 mg/dl

Exclusion Criteria:

* positive distant metastasis (including retroperitoneal lymph node metastasis)
* previous history of pelvic radiotherapy
* more than 3 months after radical surgery for cervical cancer
* neoadjuvant chemotherapy was done
* previous history of other carcinoma except for thyroid cancer, skin cancer, in situ carcinoma on cervix

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Acute toxicities according to CTCAE v4.0 | 3 months
  evaluation of acute toxicities within 3months after radiotherapy according to CTCAE v4.0

SECONDARY OUTCOMES:
Late toxicities according to CTCAE v4.0 | 5-years
  evaluation of late toxicities every year after 3months after radiotherapy according to CTCAE v4.0
Progression free survival rate | 5-years
  progression free survival rate after the time of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho WK, Park W, Kim SW, Lee KK, Ahn KJ, Choi JH. Postoperative Hypofractionated Intensity-Modulated Radiotherapy With Concurrent Chemotherapy in Cervical Cancer: The POHIM-CCRT Nonrandomized Controlled Trial. JAMA Oncol. 2024 Jun 1;10(6):737-743. doi: 10.1001/jamaoncol.2024.0565. PMID 38662364